CLINICAL TRIAL: NCT05470387
Title: A Randomized, Double-Blind, Placebo-Controlled, Study to Evaluate the Safety and Efficacy of LB1148 in Accelerating the Time to Return of Bowel Function in Subjects Undergoing Planned Bowel Resection (INTEGRITY)
Brief Title: A Study to Evaluate LB1148 for Return of Bowel Function in Subjects Undergoing Bowel Resection
Acronym: INTEGRITY
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision
Sponsor: Palisade Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PBI-POI-301
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Results first posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-04

CONDITIONS: Ileus; Gastro-Intestinal Disorder
Keywords: post operative ileus; return of bowel function; return of gastrointestinal function; enterotomy; colon surgery; colorectal surgery; intestinal surgery
MeSH Terms: conditions — Ileus; Digestive System Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LB1148 (Experimental)
  Interventions: Drug: LB1148
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LB1148 — A total of 700 mL of drug product will be administered orally as a split dose before surgery.
  Other Names: Active
  Arms: LB1148
Drug: Placebo — A total of 700 mL of placebo will be administered orally as a split dose before surgery.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of LB1148 in subjects undergoing planned bowel resection.

DETAILED DESCRIPTION:
This will be a multicenter, randomized, double-blind, placebo-controlled, study to evaluate the safety and efficacy of LB1148 in return to bowel function for subjects undergoing planned bowel resection.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for participation in the study only if they meet ALL of the following inclusion criteria:

1. Adults age 18 to 80 years, inclusive.
2. Scheduled to undergo a planned (non-emergent) bowel resection via minimally invasive technique or laparotomy. This includes any subject in which a resection of the small intestine, colon, or rectum is performed for any elective indication.
3. Willing to perform and comply with all study procedures including, being hospitalized until achieving GI-2 and responding to telephone follow-up visits as scheduled.
4. Willing and able to provide written informed consent.

Exclusion Criteria:

Subjects will not be eligible for participation in the study if they meet ANY of the following exclusion criteria:

1. History of total colectomy.
2. Has a preexisting ostomy.
3. History of radiation enteritis.
4. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2.
5. History of seizure disorder.
6. History of myeloproliferative disorders.
7. American Society of Anesthesiologists (ASA) Class IV or V.
8. Inability to take IP orally or consume solid food.
9. Planned treatment with alvimopan (Entereg®) during hospitalization period
10. Chronic opioid usage, defined by the American Pain Society as daily or near-daily use of opioids for at least 90 days.
11. Men and women of child bearing potential (WOCBP) who are unwilling to practice a highly effective method of contraception that may include, but is not limited to, abstinence, sex only with persons of the same sex, monogamous relationship with vasectomized partner, vasectomy, hysterectomy, bilateral tubal ligation, licensed hormonal methods (but not combination hormonal methods), intrauterine device, or use of spermicide combined with a barrier method (e.g., condom, diaphragm) for 28 days before Day 1 and through Day 30.
12. Women who will not agree to stop combined hormonal contraceptive and or combined hormonal replacement therapy (including combined hormonal pill, patch or vaginal ring) during the 7 day period prior to Surgery (Study Day 2) through the 7 day period following surgery (Study Days 3 through 9).
13. Has contraindications or potential risk factors to taking TXA. These include subjects with:

    * Known sensitivity to TXA
    * Recent craniotomy (past 30 days)
    * Active cerebrovascular bleed
    * Active thromboembolic disease (such as deep vein thrombosis, pulmonary embolism, cerebral thrombosis, ischemic stroke, or acute coronary syndrome)
    * Acute promyelocytic leukemia taking all-trans retinoic acid for remission induction
14. Receipt of any investigational drug within 28 days or 5 half-lives prior to Day 1.
15. Any other condition that, in the opinion of the Investigator would make the subject unsuitable for the study or unable to comply with the study requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitch Jones, MD, Study Director — CMO
Locations (23):
- United States (23):
  - Site 315, Mobile, Alabama
  - Site 354, La Jolla, California
  - Site 329, Orange, California
  - Site 350, San Diego, California
  - Site 312, Torrance, California
  - Site 359, Bridgeport, Connecticut
  - Site 351, Clearwater, Florida
  - Site 358, Jacksonville, Florida
  - Site 331, Miami, Florida
  - Site 357, Iowa City, Iowa
  - Site 321, Baltimore, Maryland
  - Site 324, Burlington, Massachusetts
  - Site 355, Grand Rapids, Michigan
  - Site 325, Rochester, Minnesota
  - Site 352, St Louis, Missouri
  - Site 317, New York, New York
  - Site 356, New York, New York
  - Site 318, Chapel Hill, North Carolina
  - Site 313, Columbus, Ohio
  - Site 353, Providence, Rhode Island
  - Site 320, Dallas, Texas
  - Site 319, Houston, Texas
  - Site 326, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- LB1148: LB1148: A total of 700 mL of drug product was administered orally as a split dose before surgery.
- Placebo: Placebo: A total of 700 mL of placebo was administered orally as a split dose before surgery.
Period: Overall Study
Arm/Group | LB1148 | Placebo
Started | 13 | 10
Completed | 13 | 7
Not Completed | 0 | 3
Not completed — Protocol Violation | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LB1148 | Placebo | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 7 | 19
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (12.59) | 54.0 (17.47) | 49.0 (15.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 9 | 5 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Time to Return of Gastrointestinal Function
Description: The later of the times in hours from placement of the last skin staple or suture to the time of toleration of solid food (defined as the time a subject finished a meal that required chewing and experienced no significant nausea/vomiting for 4 hours after the solid meal) and the first bowel movement, up to 14 days post-surgery
Time Frame: From surgical procedure up to 14 days in hospital
Population: This study was terminated early with less than 5% of the study population enrolled. As a result, formal efficacy analyses were not performed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | LB1148 | Placebo
Number analyzed (Participants) | 13 | 7
hours | 81.7 (44.67) | 90.57 (76.25)

2. Secondary Outcome: Time to First Bowel Movement
Description: Time in hours from placement of the last skin staple or suture to the time of first bowel movement
Time Frame: From surgical procedure up to 14 days in hospital
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | LB1148 | Placebo
Number analyzed (Participants) | 13 | 7
hours | 51.54 (31.08) | 46.67 (24.66)

3. Secondary Outcome: Time Subject is Ready for Discharge
Description: Time subject is ready for discharge, defined as the time from the end of surgery to the time the subject is ready for hospital discharge solely based on the recovery of GI function, as determined by the surgeon
Time Frame: From surgical procedure up to 14 days in hospital
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | LB1148 | Placebo
Number analyzed (Participants) | 13 | 7
hours | 154.48 (102.09) | 113.11 (74.75)

4. Secondary Outcome: Time Discharge Order Written
Description: Time discharge order written, defined as the time from the end of surgery to the time that the hospital discharge order is written
Time Frame: From surgical procedure up to 14 days in hospital
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | LB1148 | Placebo
Number analyzed (Participants) | 13 | 7
hours | 155.62 (100.63) | 113.11 (74.75)

5. Secondary Outcome: Time of Actual Discharge
Description: Time of actual discharge, defined as the time from the end of surgery to the time the subject is actually discharged from the hospital
Time Frame: From surgical procedure up to 14 days in hospital
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | LB1148 | Placebo
Number analyzed (Participants) | 13 | 7
hours | 159.01 (100.33) | 116.81 (75.30)

ADVERSE EVENTS:
Time Frame: All AEs were collected for all subjects during their participation from Study Day 1 through Hospital Discharge or Day 16, whichever is earlier.
Arm/Group | LB1148 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/10
Serious Adverse Events (participants affected / at risk) | 7/13 | 4/10
Other Adverse Events (participants affected / at risk) | 13/13 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LB1148 (N=13) | Placebo (N=10)
Abdominal Abscess (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anastomatic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal stoma necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic Abscess (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative Ileus (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Sepsis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LB1148 (N=13) | Placebo (N=10)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Bradycardia (Cardiac disorders) | 2 (2) | 4 (4)
Tachycardia (Cardiac disorders) | 4 (4) | 2 (2)
Visual Impairment (Eye disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural hypertension (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Procedural Hypotension (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Procedural Nausea (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperphospataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Anthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Pelvic haematoma (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT05470387/Prot_002.pdf
  • Statistical Analysis Plan (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT05470387/SAP_003.pdf